CLINICAL TRIAL: NCT00232700
Title: Investigation of Efficacy and Response Speed of a Combination Treatment of Escitalopram and Repetitive Transcranial Magnetic Stimulation
Brief Title: Investigation of a Combination Treatment of Escitalopram and rTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: H. Lundbeck A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20050041
Record Dates: First submitted 2005-10-04; First posted 2005-10-05 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2007-09

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder; Repetitive transcranial magnetic stimulation
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram

INTERVENTIONS:
Drug: Escitalopram

SUMMARY:
We intend to test in a randomized, rater blinded, placebo controlled, prospective study the primary hypothesis that an escitalopram-rTMS-combination treatment is more efficacious in the treatment of refractory major depression assessed with the Hamilton Depression Rating Scale

DETAILED DESCRIPTION:
We intend to test in a randomized, rater blinded, placebo controlled, prospective study the primary hypothesis that an escitalopram-rTMS-combination treatment is more efficacious in the treatment of refractory major depression assessed with the Hamilton Depression Rating Scale compared to placebo.

A second hypothesis is that the treatment of MDE with escitalopram (that means in the "Placebo group") alone lead to typical changes like

* An increase in neurotrophic factors concentration (measured by blood concentrations of nerve growth factor (NGF) and brain derived nerve growth factor (BDNF),
* An increase in hippocampal metabolites (measured with magnetic resonance spectroscopy (MRS
* An increase in motor cortical inhibitory activity (measured with motor evoked potentials (MEP
* An increase in serotonergic activity (measured with EEG parameters, Moreover, it is hypothesized that similar but pronounced changes occur in the group treated with the combination treatment.

ELIGIBILITY:
Inclusion Criteria:

* Major Depressive Episode (according to DSM IV standards)
* HAMD > 20
* Patient has an IQ > 70 based on the investigator´s judgement
* Patient is male or nonpregnant female adequately protected from conception
* Patient is able to comply with all testing and follow-up visit requirements defined by the study protocol
* Patient has voluntarily signed an informed consent in accordance with institutional policies

Exclusion Criteria:

* Patient has a history of schizophrenia, schizoaffective disorder or delusional disorder
* Patient currently has a secondary diagnosis of, or signs of, delirium, dementia, amnestic or other cognitive disorder per DSM IV
* Patient is suicidal
* Patient has had an alcohol or substance dependence within the previous 12 month
* Patient is currently enrolled in another investigational study
* Patient has a history of, or evidence of, significant central nervous disease (especially seizures)
* Patient has previously been treated with escitalopram
* Contraindication against escitalopram or rTMS

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2005-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of efficacy and response speed of an Escitalopram-rTMS-combination in the acute treatment of Major Depression.

SECONDARY OUTCOMES:
To determine the changes of hippocampal metabolites measured by MRS
To assess the changes of parameters of motor cortical inhibition measured by MEP
To assess the changes of NGF and BDNF
To determine the changes of event related potentials measured by electroencephalography

CONTACTS AND LOCATIONS:
Overall Officials: Malek Bajbouj, MD, Principal Investigator — Department of Psychiatry, Charité - Universitaetsmedizin Berlin, Campus Benjamin Franklin, Eschenallee 3, 14050 Berlin, Germany
Locations (1):
- Department of Psychiatry, Charité - Universitaetsmedizin Berlin, Campus Benjamin Franklin, Berlin, Germany